CLINICAL TRIAL: NCT04507997
Title: Angelman Syndrome Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: University of California, San Diego (Other); Angelman Syndrome Biomarker & Outcome Measure Consortium (A-BOM) (Unknown); Food and Drug Administration (FDA) (U.S. Federal Agency); Angelman Syndrome Foundation Canada (Unknown); Foundation for Angelman Syndrome Therapeutics Canada (Unknown); Foundation for Angelman Syndrome Therapeutics (Unknown); Angelman Syndrome Foundation, Inc. (Other)
Responsible Party: Principal Investigator, Wen-Hann Tan, Attending Physician in Genetics, Boston Children's Hospital
Other Study IDs: IRB-P00025249
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Angelman Syndrome
Keywords: Angelman syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to conduct a prospective, longitudinal natural history study of children and adults with Angelman Syndrome using investigator-observed and parent-reported outcome measures to obtain data that will be useful for future clinical trials.

DETAILED DESCRIPTION:
The overall goal is to increase our understanding of the long-term natural history of Angelman syndrome and obtain Angelman-specific norms for outcome measures that can be used in clinical trials, ultimately improving the care of individuals with Angelman syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of Angelman syndrome

Exclusion Criteria:

* Presence of another condition, unrelated to Angelman syndrome, that affects neurodevelopment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with a molecular diagnosis of Angelman syndrome
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Medical History | Through study completion, an average of 1 year
  Includes various medical complications, including seizure history
Vineland Adaptive Behavior Scales, 3rd edition | Through study completion, an average of 1 year
  Developmental and Adaptive skills
Bayley Scales of Infant and Toddler Development, 4th edition | Through study completion, an average of 1 year
  Developmental skills
Observer-Reported Communication Ability (ORCA) Measure | Through study completion, an average of 1 year
  Communication skills

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hann Tan, BMBS, Study Chair — Boston Children's Hospital
Locations (11):
- United States (8):
  - Cedars-Sinai Guerin Children's, Los Angeles, California
  - Rady Children's Hospital, San Diego, San Diego, California
  - Children's Hospital Colorado, Anschutz Medical Campus, Aurora, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - The Carolina Institute for Developmental Disabilities, Carrboro, North Carolina
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No